CLINICAL TRIAL: NCT06508346
Title: Study of Therapeutic Efficacy of Anti-CD19 CAR-T Cells in Children With Refractory ANCA-Associated Vasculitis
Brief Title: Study of Therapeutic Efficacy of Anti-CD19 CAR-T Cells in Children With Refractory Refractory AAV
Status: Recruiting | Type: Observational
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Mao Jianhua, professor, The Children's Hospital of Zhejiang University School of Medicine
Other Study IDs: 2024-IRB-0163-P-01
Record Dates: First submitted 2024-07-14; First posted 2024-07-18 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: ANCA Associated Vasculitis; CAR-T Cell Therapy
Keywords: AAV; ANCA Associated Vasculitis; CAR-T cell therapy
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: anti-CD19-CAR-T cells — Intravenous injection

SUMMARY:
This is an investigator-initiated trial aimed at assessing the safety and efficacy of anti-CD19 CAR-T cells in the treatment of childhood-onset refractory ANCA-Associated Vasculitis.

DETAILED DESCRIPTION:
The anti-neutrophil cytoplasmic antibody (ANCA) associated vasculitis （AAV ）is one of the most devastating and potentially fatal autoimmune diseases, characterized by involvement of small blood vessels (arterioles, tiny arteries, tiny static veins, and capillaries) and the presence of ANCA. The disease lead to extensive damage in multiple organs and systems,such as pulmonary hemorrhage and rapidly progressive glomerulonephritis (RPGN),ultimately resulting in disability and even death.Children with AAV are particularly at risk of organ damage, especially to the kidneys, and tend to more serious than that in adults.

Currently, the primary treatment for AAV relies on glucocorticoids and immunosuppressants to alleviate symptoms. However, due to the absence of a curative treatment, patients often require lifelong medication. In recent years, biological agents such as rituximab have been introduced for the treatment of AAV, but still cannot completely eliminate autoimmune B cells in the bone marrow, leading to unsatisfactory overall outcomes. Furthermore, stopping the drugs can lead to relapse, and there is still no cure for AAV, leaving patients facing the challenges of lifelong medication and an incurable disease.

Since 2019, CAR-T cell therapy has been successfully applied to autoimmune diseases. Clinical studies have demonstrated that targeted CD19 CAR-T cells hold significant therapeutic potential for SLE. These cells effectively slow down the pathological progression of SLE and can also effectively treat severe cases. Furthermore, targeted CD19 CAR-T cells are also expected to restore the immune system in SLE patients, potentially allowing them to discontinue lifelong medication and avoid serious long-term side effects of drugs like hormones and immunosuppressants. Studies have reported that CAR-T has a good therapeutic effect on a variety of autoimmune diseases such as systemic sclerosis and idiopathic inflammatory dermatomyositis.The purpose of this study is to assess the safety and efficacy of the anti-CD19 CAR-T cells in the treatment of childhood-onset refractory AAV.

ELIGIBILITY:
Inclusion Criteria:

1. Age:5-25 years old(including threshold);
2. Diagnosed with AAV according to the 2022EULAR/ACR AAV classification criteria；despite of the Treatment with glucocorticoids (more than 1mg/kg/ day), cyclophosphamide, and rituximab for at least 3 months, still cannot achieve sustained response or disease recurred after response; Or use glucocorticoid combined with cyclophosphamide/rituximab plus more than one of the other immunosuppressants (including azathioprine, moxophenolate, methotrexate, leflunomide, tacrolimus, cyclosporine, beliuzumab, etc.) ≥3months，still failed to achieve sustained remission or relapsed after remission; Or meet the diagnostic criteria for severe vasculitis, clinical routine treatment is ineffective, the benefit is judged by the investigator to outweigh the risk, and the patient or guardian has fully informed consent, can be considered for inclusion。
3. patient <18 years old：PVAS≥15（total 63）；≥18 years old: BVAS≥15(total 63)
4. The functions of important organs are basically normal: Cardiac function: Left ventricular ejection fraction (LVEF) ≥55% with no obvious abnormality in electrocardiogram; Renal function: eGFR≥30ML/min/1.73m2； Liver function: Asparagus cochinchinensis transase (AST) and Alanine Aminotransferase (ALT)≤3.0 ULN, Total Bilirubin (TBIL) in serum ≤2.0×ULN; Lung function: No serious lung lesions, SpO2≥92%;
5. Met the standards of leukapheresis or intravenous blood collection, No contraindication for cell collection;
6. Negative pregnancy test for female Subjects of childbearing age, agree to take effective contraceptive measures the first year after CAR-T infusion;
7. Participants or their guardians agrees to participate in the clinical trial and sign the informed consent form which indicating that he/she understands the purpose and procedure of the clinical trial and is willing to participate in the study.

Exclusion Criteria:

1. Received CAR T cell therapy previously;
2. Central nervous system (CNS) disease: CNS neurolupus requires intervention within 60 days);
3. Pulmonary hemorrhage that need for pulmonary ventilation support for more than 1 week;
4. Have a history of congenital heart disease or acute myocardial infarction within 6 months prior to screening; Or severe arrhythmias (including multisource frequent supraventricular tachycardia, ventricular tachycardia, etc.); Or combined with moderate to massive pericardial effusion, serious myocarditis, etc; Or patients with unstable vital signs who need hypertensive drugs；
5. Suffer from other diseases that require long-term use of glucocorticoid or high-dose of immunosuppressive agents;
6. Uncontrollable infection, or active infection that requires systemic treatment within 1 week prior to screening；
7. History of organ transplantation or hematopoietic stem cell transplantation, or ≥Grade 2 GVHD within 2 weeks prior to screening；
8. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer greater than the normal reference value range; Or hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA titer greater than the normal reference value range; Or positive for human immunodeficiency virus (HIV) antibodies; Or syphilis test positive; Or cytomegalovirus (CMV) DNA test positive;
9. Received live vaccine within 4 weeks before screening;
10. Tested positive in Blood pregnancy test；
11. Previous or concurrent malignancy；
12. Patients who participated in other clinical study within 3 months prior to enrollment;
13. Any other conditions that the investigators deem it unsuitable for the study

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The trial consists of two phases, Dose Exploration (Part A) and Dose Expansion (Part B). In Part A, two dose groups (0.3×10^5/kg, 1×10^5/kg,) are set up, starting from the low dose group to explore the safe and effective dose. If the optimal effective dose is still not explored in the highest dose group, the dose can be increased according to the situation, and the highest dose is no more than 3×10^5/kg. Upon the completion of Part A, the optimal dose is selected by the comprehensive judgment of the investigator and the technical partner to enter into the Part B stage. with this dose , anther 3 cases are enrolled to continue to validate the safety and efficacy. A total enrollment of 9-12 patients is expected in the whole process of the trial.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The safety of CAR-T cell in refractory childhood-onset ANCA-Associated Vasculitis | 3 months and 6 months
  The number of occurrence and proportion of adverse events and serious adverse events that occurred

SECONDARY OUTCOMES:
The efficiency of CAR-T cell in refractory childhood-onset AAV | 3 months and 6 months
  Percentage of patients achieving 50% response 100% response by the 3-month time
The efficiency of CAR-T cell in refractory childhood-onset AAV | 3 months
  the assessment of disease activity using PVAS/BVAS 3.0 ,the asseeement of the Irreversible damage by PVDI/VDI,and the changes in laboratory values
Cellular kinetics | 6 months
  CAR transgene levels by quantitative polymerase chain reaction (qPCR) in peripheral blood.
Autoantibody detection | 24 months
  Autoantibody detection up after CD19 CAR-T cells infusion.
Duration of disease response (DOR) | 24 months
  the time between the first investigator assessment of remission and the first investigator assessment of progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Mao, PhD, Principal Investigator — Children's Hospital, Zhejiang University School of Medicine; Mo Wang, PhD, Principal Investigator — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No